CLINICAL TRIAL: NCT01472185
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Ranolazine Monotherapy in Subjects With Type 2 Diabetes Mellitus
Brief Title: Ranolazine Monotherapy in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-259-0131
Record Dates: First submitted 2011-11-11; First posted 2011-11-16 (Estimated); Results first posted 2014-10-15 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ranolazine; Diet; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Qualifying Period: Placebo to match ranolazine (1 tablet twice daily) for 14 days.
  Treatment Period: Placebo to match ranolazine (Days 1-7: 1 tablet twice daily; 2 tablets twice daily thereafter) for up to 24 weeks.
  Participants were required to maintain their diet and exercise regimen.
  Interventions: Drug: Placebo; Behavioral: Diet; Behavioral: Exercise
- Ranolazine (Experimental): Qualifying Period: Placebo to match ranolazine (1 tablet twice daily) for 14 days.
  Treatment Period: Ranolazine tablets (Days 1-7: 1 × 500 mg twice daily; 2 × 500 mg twice daily thereafter) for up to 24 weeks.
  Participants were required to maintain their diet and exercise regimen.
  Interventions: Drug: Ranolazine; Drug: Placebo; Behavioral: Diet; Behavioral: Exercise

INTERVENTIONS:
Drug: Ranolazine — Ranolazine tablets administered orally twice daily.
  Other Names: Ranexa®
  Arms: Ranolazine
Drug: Placebo — Placebo to match ranolazine administered orally twice daily.
Behavioral: Diet — Participants are instructed to continue the diet regimen prescribed by their physician.
Behavioral: Exercise — Participants are instructed to continue the exercise regimen prescribed by their physician.

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group, multi-center study to determine the effect of ranolazine when given as monotherapy on glycemic control in subjects with type 2 diabetes mellitus (T2DM) who were inadequately controlled with diet and exercise alone and who are treatment naive to antihyperglycemic therapy or have not received antihyperglycemic therapy in the 90 days (or thiazolidinediones [TZDs] for at least 24 weeks) prior to screening, and to characterize the relationship between HbA1c reduction and other glycemic parameters in subjects with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Males and females, 18 to 75 years old, inclusive
* Documented history of T2DM
* Treatment naïve to antihyperglycemic therapy or having received no prior treatment with antihyperglycemic therapy for at least 90 days (TZDs for at least 24 weeks) prior to screening
* Body mass index (BMI) 25 kg/m2 to 45 kg/m2 inclusive at screening
* HbA1c 7% - 10%, inclusive at screening and at the end of the Qualifying Period (Day 14 +2 days)
* Fasting serum glucose (FSG) of ≥ 130 mg/dL (7.2 mmol/L) and ≤ 240 mg/dL (13.3 mmol/L) at screening and at the end of the Qualifying Period (Day 14 +2 days). A one-time central laboratory re-test of FSG is allowed in subjects with an initial central laboratory FSG ≥ 125 mg/dL (6.9 mmol/L) and < 130 mg/dL (7.2 mmol/L) who are otherwise eligible as determined by the investigator.
* Fasting serum C-peptide ≥ 0.8 ng/mL at screening
* Able and willing to comply with all study procedures during the course of the study
* Females of child-bearing potential must have a negative pregnancy test at screening and must agree to use highly effective contraception methods from screening throughout the duration of the Treatment Period and for 14 days following the last dose of study drug
* At least 80% compliant with dosing during the Qualifying Period

Exclusion Criteria:

* History of or current diagnosis of type 1 diabetes mellitus
* History of diabetic ketoacidosis, ketosis-prone diabetes, or hyperosmolar hyperglycemic coma
* History of a severe episode of hypoglycemia (≥ 1 episode within 3 months prior to screening or ≥ 2 episodes within 6 months prior to screening), defined as hypoglycemia requiring 3rd party assistance to actively administer carbohydrate, glucagon, or other resuscitative actions due to severe impairment in consciousness or behavior
* Clinically significant complications of diabetes that, in the judgment of the investigator, would make the subject unsuitable to participate in this study
* History of any clinically significant cardiovascular or cerebrovascular event (eg, myocardial infarction [MI], acute coronary syndrome [ACS], recent coronary revascularization [including coronary artery bypass graft procedures or percutaneous coronary intervention], transient ischemic attack or ischemic stroke) ≤ 3 months prior to screening
* Inadequately controlled or unstable hypertension as defined by systolic blood pressure (SBP) > 160 mmHg or diastolic blood pressure (DBP) > 100 mmHg at screening and randomization
* Prolonged QTc interval > 500 msec by ECG at screening, a personal or family history of QTc prolongation, congenital long QT syndrome, or subjects who are receiving drugs that prolong the QTc interval, such as Class Ia or Class III antiarrhythmic agents, erythromycin, and certain antipsychotics (eg, ziprasidone)
* History of bariatric surgery at any time in the past or any other surgery < 2 months before screening, or planning to undergo surgery during the study. Subjects with a planned minor surgery may be enrolled upon approval by the Medical Monitor.
* Any other hospitalization in the 14 days prior to screening or planned hospitalization at any time during the study
* Significant weight change (± 5%) < 2 months prior to screening or on a weight-loss program and is not in the maintenance phase at screening
* Severe renal impairment, defined as an estimated glomerular filtration rate (eGFR) by the Modification of Diet in Renal Disease (MDRD) equation < 30 mL/min/1.73 m2 at screening or undergoing any type of dialysis at screening or planning to undergo any type of dialysis during the course of the study.
* History of liver cirrhosis (Child-Pugh Class A, B or C)
* Active liver disease and/or significant abnormal liver function defined as aspartate aminotransferase (AST) > 3x upper limit of the normal range (ULN) and/or alanine aminotransferase (ALT) > 3x ULN and/or serum total bilirubin > 2.0 mg/dL
* History of cancer (except non-melanomic skin cancers or cervical in situ) within 5 years prior to screening
* History of alcohol or other drug abuse < 12 months prior to screening
* Any other clinically significant existing medical or psychiatric condition, including clinically significant laboratory abnormalities, or one requiring further evaluation that, in the opinion of the investigator, could interfere with conduct of the study or interpretation of the data
* Prior treatment with open-label ranolazine or known hypersensitivity or intolerance to ranolazine or any of its excipients
* Treatment with strong or moderate cytochrome (CYP)3A inhibitors or P-glycoprotein (P-gp) inhibitors within 14 days prior to randomization
* Treatment with CYP3A inducers or P-gp inducers within 14 days prior to randomization
* Treatment with CYP3A4 substrates with a narrow therapeutic range (eg, cyclosporine, tacrolimus, sirolimus) within 14 days prior to randomization
* Treatment with simvastatin at a daily dose > 20 mg or lovastatin at a daily dose > 40 mg, within 14 days prior to randomization
* Weight-loss medication or anti-obesity medication (prescription or nonprescription) < 3 months prior to screening
* Treatment with niacin > 200 mg daily; if receiving ≤ 200 mg daily, should be on stable doses for ≥ 90 days prior to screening and for the duration of the study
* Expected or current treatment with systemic corticosteroids (oral or injectable) for > 14 days from screening through the end of the Treatment Period. Topical or inhaled corticosteroid formulations are permitted at any time during the study
* If receiving thyroid replacement therapy, should be on stable doses for at least 6 weeks prior to randomization
* Hemoglobin < 12 g/dL for males; or < 11 g/dL for females, at screening
* Participation in another clinical study involving an investigational drug or device < 30 days prior to screening; participation in another clinical study involving an antihyperglycemic therapy < 90 days prior to screening
* Donation of blood < 2 months prior to screening; plans to donate blood while participating in the study
* Females who are pregnant or breastfeeding
* Other condition(s) that, in the opinion of the investigator, would compromise the safety of the subject, would prevent compliance with the study protocol (including the ability to comply with Mixed Meal Tolerance Test [MMTT]), or would compromise the quality of the clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2011-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (158):
- United States (57):
  - Thunderbird Internal Medicine/Clinical Research Advantage, Glendale, Arizona
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Desert Sun Clinical Research, LLC, Tucson, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - North Central Arkansas Medical Associates, Mountain Home, Arkansas
  - Paul W. Davis, MD, Private Practice, Pine Bluff, Arkansas
  - Southland Clinical Research Center, Inc., Fountain Valley, California
  - Global Research Management, Glendale, California
  - National Research Institute, Los Angeles, California
  - Spectrum Clinical Research Institute, Inc, Moreno Valley, California
  - Sacramento Heart and Vascular Medical Associates, Sacramento, California
  - Clearview Medical Research LLC, Santa Clarita, California
  - Infosphere Clinical Research, West Hills, California
  - Boca Raton Clinical Research Associates, Inc, Boca Raton, Florida
  - PAB Clinical Research, Brandon, Florida
  - Florida Research Network, LLC, Gainesville, Florida
  - A G A Clinical Trials, Hialeah, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Baptist Diabetes Associates, Miami, Florida
  - NextPhase Clinical Trials, Inc., Miami Beach, Florida
  - Precision Research Organization, Miami Lakes, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Florida Institute for Clinical Research LLC, Orlando, Florida
  - Regenerate Clinical Trials, South Miami, Florida
  - Synergy Therapeutic Partners, Atlanta, Georgia
  - CTL Research, Eagle, Idaho
  - Cedar-Crosse Research Center, Chicago, Illinois
  - LaPorte County Institute for Clinical Research, Michigan City, Indiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - MD Medical Research, Oxon Hill, Maryland
  - IRC Clinics, Inc, Towson, Maryland
  - Associated Internal Medicine Specialists, P.C., Battle Creek, Michigan
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - University of New Mexico Clinical and Translational Science Center, Albuquerque, New Mexico
  - Clinical Research Solution, New York, New York
  - PMG Research of Charlotte, Charlotte, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Clinical Inquest Center, Ltd., Beavercreek, Ohio
  - Infinity Research Group, LLC, Oklahoma City, Oklahoma
  - Blair Medical Associates, Inc, Station Medical Center, Altoona, Pennsylvania
  - Southeastern Research Associates, Inc., Taylors, South Carolina
  - HCCA Clinical Research Solutions, Columbia, Tennessee
  - HCCA Clinical Research Solution, Jackson, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - HCCA Clinical Research Solutions, Smyrrna, Tennessee
  - The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Excel Clinical Research, LLC, Houston, Texas
  - Texas Center for Drug Development, PA, Houston, Texas
  - Humble Cardiology Associates, Humble, Texas
  - Juno Research, LLC, Katy, Texas
  - Cetero Research, San Antonio, Texas
  - Discovery Clinical Trials, San Antonio, Texas
  - Highland Clinical Research, Salt Lake City, Utah
  - Jean Brown Research, Salt Lake City, Utah
  - Burke Internal Medicine & Research, Burke, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
- Nemocnice s poliklinikou Havirov, Havířov, Moravskoslezský kraj, Czechia
- Hungary (7):
  - Drug Research Center, Balatonfüred
  - Synexus Hungary Ltd, Budapest
  - Markhot Ferenc Hospital, Eger
  - Kanizsai Dorottya Hospital, Nagykanizsa
  - Borbanya Praxis Kft., Outpatient Clinic, Nyíregyháza
  - Medifarma 98, Nyíregyháza
  - Zala County Hospital, Zalaegerszeg
- Poland (14):
  - LANDA - Specjalistyczne Gabinety Lekarskie, Krakow, Lesser Poland Voivodeship
  - NZOZ Centrum Badan Klinicznych Oswiecim, Oswięcim, Lesser Poland Voivodeship
  - NZOZ Regionalna Poradnia Diabetologiczna, Wroclaw, Lower Silesian Voivodeship
  - NZOZ Centrum Badan Klinicznych, Wroclaw, Lower Silesian Voivodeship
  - NZOZ Centrum Osteporozy i Chorob Kostno-Stawowych J.Badurski Sp.j., Bialystok
  - Leszek Romanowski Barbara Romanowska "DIABET" Centrum Medyczne s.c., Chrzanów
  - NZOZ Specjalistyczna Przychodnia Medyczna Atopia, Krakow
  - NZOZ Cereo-Med Sp. z o.o., Lodz
  - Specjalistyzny Ośrodek Lecznicz-Badawczy, Ostróda
  - Miedzyleski Szpital Specjalistyczny w Warszawie, Warsaw
  - SPZOZ Uniwersytecki Szpital Kliniczny Nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Łodzi, Oddział Kliniczny Diabetologii, Lodz, Łódź Voivodeship
  - NZOZ Centrum Medyczne Szpital Sw. Rodziny, Lodz, Łódź Voivodeship
  - NZOZ Polimedica, Zgierz, Łódź Voivodeship
  - NZOZ PrimaMED, Kielce, Świętokrzyskie Voivodeship
- Romania (11):
  - CMI Morosanu V. Magdalena, Galati, Galați County
  - Spitalul Clinic Judetean de Urgenta "Sf. Apostol Andrei" Galati, Galati, Galați County
  - Spital Clinic Judetean de Urgenta Oradea Stationarul 1, Oradea, Jud Bihor
  - Vitadiab SRL - Cabinet Medical Dr. Barabas Alina SRL, Brasov, Jud Brasov
  - Consultmed SRL, Iași, Jud. Iasi
  - CMI Diabet Nutritie Boli Metabolice Dr. Pop Lavinia, Baia Mare, Jud. Maramures
  - Diabmed Dr. Popescu Alexandrina SRL, Ploieşti, Prahova
  - Institutul de Diabet, Nutritie si Boli Metabolice "Dr. N. C. Paulescu", Bucharest
  - Tehnomed Trading Srl, Bucharest
  - O.D. Medica Srl, Bucharest
  - Centru Medical Dr. Negrisanu, Timisoara, Jud. Timis
- Russia (38):
  - 3rd Central Military Clinical Hospital named after A.A.Vishnevskogo, Arkhangel'skoye
  - GOU VPO "Chita State Medical Academy" of Minzdravsocrazvitie RF, Chita
  - "Clinic of New Medical Technology" Company Limited, Dzerzhinskiy
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - "Krasnoyarsk State Medical University n.a. Prof. V.F. Voyno-Yasenetsky, Krasnoyarsk
  - State Healthcare Institution of Moscow "Cardiologival Dispensary #2 of Management Department of South Administrative District", Moscow
  - Central Clinical Hospital of Russian Academy of Sciences, Moscow
  - Medical Sanitary Unit of Minestry of Internal Affairs of Russia in Moscow, Moscow
  - Moscow City Clinical Hospital #63, Moscow
  - City Clinical Hospital # 13 of Avtozavodsky District of Nizhniy Novgorod, Nizhny Novgorod
  - Novosibirsk State Medical University, Novosibirsk
  - LLC "Reafan", Novosibirsk
  - Scientific Research Institute of Physiology of Siberian Department RAMS, Novosibirsk
  - City Hospital # 38 named after N A Semashko, Pushkin
  - Rostov State Medical University, Rostov-on-Don
  - Ryazan State Medical University, Ryazan
  - Saint-Petersburg City Outpatient Clinic#37, Saint Petersburg
  - Medinet, LLC, Saint Petersburg
  - North-Western State Medical Unversity n.a. I.I.Mechnikov, Saint Petersburg
  - Military Medical Academy named after S.M. Kirov, Saint Petersburg
  - Saint-Petersburg state budgetary healthcare institution "City Polyclinic #109", Saint Petersburg
  - Alexanders City Hospital, Saint Petersburg
  - Clinical Hospital #122 n.a. Sokolov of FMBA, Saint Petersburg
  - ANO "Medical Centre "XXI century", Saint Petersburg
  - St. Elizabeth City Hospital, Saint Petersburg
  - Krestovsky Island Medical Institute, LLC, Saint Petersburg
  - Federal Centre of Heart, Blood and Endocrinology named after V.A. Almazov, Saint Petersburg
  - International Medical Center "SOGAZ", LLC, Saint Petersburg
  - Saint-Petersburg City Pokrovskaya Hospital, Saint Petersburg
  - Center "Diabetes", LLC, Samara
  - Smolensk State Medical Academy, Sanatorium-Preventorium, Smolensk
  - Tyumen State Medical Academy, Tyumen
  - Voronezh Regional Clinical Hospital #1, Voronezh
  - City Hospital named after N.A.Semashko, Yaroslavl
  - Clinical Hospital for Emergency Care named after N.V. Solovyov, Yaroslavl
  - Medical Sanitary Unit of Novo-Yaroslavsky Oil Refinery, Yaroslavl
  - Yaroslavl Regional Clinical Hospital, Yaroslavl
  - The Urals State Medical Academy, Yekaterinburg
- Serbia (2):
  - Clinical Center of Serbia, Belgrade
  - Clinical Center of Kragujevac, Kragujevac
- Slovakia (7):
  - METABOLKLINIK s.r.o., Bratislava, Bratislava Region
  - Metabolic Center of Dr. Katarina Raslova Ltd., Bratislava, Bratislava Region
  - "Diabetologicka a metabolicka ambulancia Human-care s.r.o", Košice, Košice Region
  - ARETEUS s.r.o., Diabetologicka ambulancia, Trebišov, Košice Region
  - MediVet s.r.o., Malacky
  - ENDIAMED s.r.o, Dolný Kubín, Žilina Region
  - MEDIVASA s.r.o., Žilina, Žilina Region
- South Africa (9):
  - Newkwa Medical Centre, Newlands West, Durban
  - Global Clinical Trials, Pretoria, Pretoria
  - Netcare Umhlanga Medical Centre, Kwa Zulu Natal, Umhlanga, Durban
  - Worthwhile Clinical Trials, Benoni
  - Centre for Diabetes, Asthma and Allergy, Johannesburg
  - Soweto Clinical Trial Centre, Johannesburg
  - Aliwal Shoal Medical & Clinical Trial Centre, Kwa Zulu Natal
  - Helderberg Clinical Trials Centre, Somerset West
  - Tiervlei Trial Centre, Western Cape
- Ukraine (12):
  - City Clinical Hospital#9, Dnipropetrovsk State Medical Academy, Dnipropetrovsk
  - Educational Scientific Medical Centre "University clinic" of Donetsk National Medical University n.a. M.Gorkiy, Donetsk
  - State Institution "Institute of Problems of Endocrine Pathology n.a. V.Y. Danylevsky of NAMS of Ukraine", Kharkiv
  - Administration of Medical Service and Rehabilitation of "ARTEM" State Holding Company, Kyiv
  - National Medical University n.a. O.O. Bogomolets, Chair of Family Medicine based on Outpatient Clinic # 2 of Shevchenkovsky District, Kyiv
  - V. P. Komissarenko Institute of Endocrinology and Metabolism of AMS of Ukraine, Kyiv
  - Municipal Institution Lutsk City Clinical Hospital, Lutsk
  - Lviv Regional Endocrinology Dispensary, Lviv
  - Odessa State Medical University, Odesa
  - Public Institution "City Outpatients' Hospital #20", Odesa
  - Vinnytsya Regional Clinical Endocrinology Dispensary, Vinnytsia
  - Zhytomyr Regional Clinical Hospital, Zhytomyr

REFERENCES:
- [Derived] Eckel RH, Henry RR, Yue P, Dhalla A, Wong P, Jochelson P, Belardinelli L, Skyler JS. Effect of Ranolazine Monotherapy on Glycemic Control in Subjects With Type 2 Diabetes. Diabetes Care. 2015 Jul;38(7):1189-96. doi: 10.2337/dc14-2629. Epub 2015 Jun 6. PMID 26049552

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 113 study sites in the United States, South Africa, Europe, and Russia. The first participant was screened on 15 November 2011. The last participant observation occurred on 21 October 2013.
Pre-assignment Details: 605 participants entered the qualifying period; 465 were randomized, and 464 were randomized and treated (Safety Analysis Set). Of these, 8 were excluded due to major eligibility criteria protocol violation or had baseline but no on-treatment data; thus, 456 were included in the Full Analysis Set.
Period: Overall Study
Arm/Group | Placebo | Ranolazine
Started | 232 | 233
Completed | 198 | 199
Not Completed | 34 | 34
Not completed — Randomized but Not Treated | 0 | 1
Not completed — Adverse Event Other than Hyperglycemia | 3 | 10
Not completed — Hyperglycemia | 5 | 2
Not completed — Investigator's Discretion | 3 | 1
Not completed — Lost to Follow-up | 4 | 1
Not completed — Protocol Violation | 5 | 1
Not completed — Subject Noncompliance | 8 | 15
Not completed — Subject Withdrew Consent | 6 | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for the Safety Analysis Set following randomization. The Safety Analysis Set includes randomized participants who received at least one dose of study treatment, analyzed based on actual treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ranolazine | Total
Number analyzed (Participants) | 232 | 232 | 464
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (9.3) | 55 (9.5) | 56 (9.4)
Age, Customized [Number; unit: participants]
  < 65 years | 197 | 199 | 396
  ≥ 65 years | 35 | 33 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 123 | 236
  Male | 119 | 109 | 228
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 29 | 60
  Not Hispanic or Latino | 201 | 202 | 403
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 10 | 9 | 19
  Black or African-American | 10 | 9 | 19
  White | 209 | 213 | 422
  Other | 2 | 1 | 3
  Not Permitted | 1 | 0 | 1
Region of Enrollment [Number; unit: participants] — All randomized participants were analyzed for region of enrollment (placebo, n = 232; ranolazine, n = 233).
  participants
    Serbia | 0 | 2 | 2
    United States | 62 | 56 | 118
    Hungary | 12 | 9 | 21
    Slovakia | 8 | 13 | 21
    Poland | 7 | 11 | 18
    Ukraine | 39 | 36 | 75
    Romania | 10 | 11 | 21
    South Africa | 11 | 13 | 24
    Russian Federation | 83 | 82 | 165
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.8 (4.85) | 32.8 (4.75) | 32.8 (4.80)
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent HbA1c in blood] | 8.01 (0.727) | 8.06 (0.732) | 8.04 (0.729)
Fasting Serum Glucose [Mean (Standard Deviation); unit: mg/dL] | 171.5 (34.45) | 172.1 (34.32) | 171.8 (34.35)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 3.0 (4.00) | 3.0 (4.29) | 3.0 (4.14)
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 83.3 (18.40) | 84.5 (18.80) | 83.9 (18.59)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: The average (mean) change from baseline in HbA1c at Week 24 was analyzed.
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set (randomized participants who received ≥ 1 dose of study treatment with a baseline and at least one postbaseline measurement of HbA1c, excluding subjects with major eligibility violations and analyzed based on the randomized treatment regardless of actual treatment received) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent of HbA1c in blood
Arm/Group | Placebo | Ranolazine
Number analyzed (Participants) | 195 | 199
percent of HbA1c in blood
  HbA1c at Week 24 | 7.70 (1.183) | 7.26 (1.101)
  Change from baseline in HbA1c at Week 24 | -0.27 (1.027) | -0.80 (1.020)
Statistical Analysis 1: Comparison: Placebo vs Ranolazine; Assuming a common standard deviation of 1.2%, an effective sample size of 400 would provide at least 90% power to detect a statistically significant treatment difference of -0.5% (ranolazine vs. placebo) for the reduction of HbA1c from baseline at Week 24 based on a 2-sided alpha of 0.05 and 1:1 randomization; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model Analysis — P-value is from a mixed effects model including terms for baseline HbA1c value, treatment group, visit week, and treatment by visit week interaction. Unstructured covariance matrix was used; difference in least squares mean (LSM) = -0.56, 95% CI 2-sided [-0.76 to -0.36] — The estimation (LSM) is of the placebo-corrected change from baseline

2. Secondary Outcome: Change From Baseline in Fasting Serum Glucose at Week 24
Description: The average (mean) change from baseline in fasting serum glucose at Week 24 was analyzed.
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Ranolazine
Number analyzed (Participants) | 191 | 197
mg/dL | 1 (42.2) | -7 (37.5)

3. Secondary Outcome: Percentage of Participants With HbA1c < 7% at Week 24
Time Frame: Week 24
Population: Participants in the Full Analysis Set with Baseline HbA1c ≥ 7% and available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ranolazine
Number analyzed (Participants) | 195 | 199
percentage of participants | 25.6 | 41.2

4. Secondary Outcome: Change From Baseline in 2-hour Postprandial Serum Glucose at Week 24
Description: The average (mean) change from baseline in 2-hour postprandial serum glucose at Week 24 was analyzed.
  Mixed Meal Tolerance Test (MMTT) Full Analysis Set: randomized participants who received at least one dose of study treatment with a baseline and at least one postbaseline measurement of serum glucose at time [T] = 120 minutes during the MMTT, administered under fasting conditions, excluding participants with major eligibility protocol violations and analyzed based on the randomized treatment regardless of actual treatment received.
Time Frame: Baseline; Week 24
Population: Participants in the Mixed Meal Tolerance Test (MMTT) Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Ranolazine
Number analyzed (Participants) | 178 | 185
mg/dL | 2 (65.1) | -19 (53.8)

5. Secondary Outcome: Change From Baseline in Incremental Change of 2-hour Postprandial Serum Glucose at Week 24
Description: The average (mean) change from baseline in incremental change of 2-hour postprandial serum glucose at Week 24 was analyzed.
Time Frame: Baseline; Week 24
Population: Participants in the Mixed Meal Tolerance Test (MMTT) Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Ranolazine
Number analyzed (Participants) | 173 | 180
mg/dL | -1 (47.7) | -12 (37.9)

ADVERSE EVENTS:
Time Frame: Up to 24 Weeks plus 30 days
Description: Safety Analysis Set: randomized participants who received at least one dose of study treatment, analyzed based on actual treatment received.
Arm/Group | Placebo | Ranolazine
Serious Adverse Events (participants affected / at risk) | 7/232 | 6/232
Other Adverse Events (participants affected / at risk) | 31/232 | 28/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=232) | Ranolazine (N=232)
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Sinoatrial block (Cardiac disorders) | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Non-small cell lung cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=232) | Ranolazine (N=232)
Hyperglycaemia (Metabolism and nutrition disorders) | 23 | 18
Headache (Nervous system disorders) | 10 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years